CLINICAL TRIAL: NCT01827592
Title: A Double-blind, Randomised, Placebo-controlled, Phase 3 Trial in Patients With Chronic Idiopathic Constipation to Demonstrate the Efficacy and Safety of Elobixibat 5 mg and 10 mg for 26 Weeks
Brief Title: 26 Week Efficacy and Safety Trial for Patients With Chronic Idiopathic Constipation
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated due to a distribution issue with the trial medication
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 000079; 2012-005587-94 (EudraCT Number)
Record Dates: First submitted 2013-04-05; First posted 2013-04-09 (Estimated); Results first posted 2015-10-20 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-09

CONDITIONS: Chronic Idiopathic Constipation
MeSH Terms: interventions — elobixibat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- EBX 10 (Experimental): Elobixibat 10 mg/day
  Interventions: Drug: Elobixibat 10 mg
- EBX 5 (Experimental): Elobixibat 5 mg/day
  Interventions: Drug: Elobixibat 5 mg
- PLCBO (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Elobixibat 10 mg — Elobixibat 10 mg/day
  Other Names: A3309
  Arms: EBX 10
Drug: Elobixibat 5 mg — Elobixibat 5 mg/day
  Other Names: A3309
  Arms: EBX 5
Drug: Placebo — Placebo
  Arms: PLCBO

SUMMARY:
Efficacy and Safety Trial of elobixibat in Patients with Chronic Idiopathic Constipation treated for 26 Weeks.

DETAILED DESCRIPTION:
The present trial was designed to determine the efficacy and safety of elobixibat treatment (at both doses of 5 mg and 10 mg/day) compared to placebo treatment for 26-week Treatment Period in patients with chronic idiopathic constipation. Patients were followed-up for 2 weeks after end of the Treatment Period.

The assessment of primary and key secondary end points was done for patients who completed the first 12 weeks of Treatment Period. Incidence of Adverse Events (AEs) were reported till 2 weeks after end of the treatment.

The trial was early terminated due to a distribution issue with the trial medication.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) ≥18.5 but <35.0 kg/m^2
* Male or female ≥18 years of age
* Reports <3 spontaneous Bowel movements (BM) per week and reports one or more of the following symptoms for the last 3 months with symptom onset at least 6 months before the Screening Visit or before starting chronic therapy with any laxative:

  1. Straining during at least 25% of defecations
  2. Lumpy or hard stools during at least 25% of defecations
  3. Sensation of incomplete evacuation during at least 25% of defecations
* Is ambulatory and community dwelling
* An initial colonoscopy is required if recommended by national guidelines

Exclusion Criteria:

* Reports loose (mushy) or watery stools in the absence of any laxative intake in the form of a tablet, a suppository or an enema, or prohibited medicine for >25% of BMs
* The patient reports a BSFS of 6 or 7 during the Pretreatment Period
* Has irritable bowel syndrome (IBS) with pain/discomfort as predominant symptoms
* Has a structural abnormality of the GI tract or a disease or condition that can affect Gastrointestinal (GI) motility
* Has a history of diverticulitis, chronic pancreatitis, active peptic ulcer disease (PUD) not adequately treated, ischaemic colitis, inflammatory bowel disease, laxative abuse, faecal impaction that required hospitalization or emergency treatment, pseudo-obstruction, megacolon, megarectum, bowel obstruction, descending perineum syndrome, ovarian cysts, endometriosis, solitary rectal ulcer syndrome, systemic sclerosis, pre-malignant colonic disease (e.g., familial adenomatous polyposis or hereditary non-polyposis colorectal cancer) or other forms of familial colorectal cancer.
* Has unexplained and clinically significant GI alarm signals (e.g., lower GI bleeding or heme-positive stool in the absence of known internal or external haemorrhoids, iron-deficiency anaemia, unexplained weight loss) or systemic signs of infection or colitis
* Has a potential central nervous system (CNS) cause of constipation (e.g., Parkinson's disease, spinal cord injury, multiple sclerosis)
* Has intestinal/rectal prolapse or other known pelvic floor dysfunction
* Commonly uses digital manoeuvres (perianal pressure or digital disimpaction) or vaginal splinting to facilitate the passage of a bowel movement
* Has a history of diabetic neuropathy
* Has a history of bariatric surgery for treatment of obesity; surgery to remove a segment of the GI tract; or surgery of the abdomen, pelvic or retroperitoneal area during the 6 months prior to Screening; or appendectomy or cholecystectomy 3 months prior to screening; or other major surgery 1 month prior to Screening
* Has a history of cancer with last date of proven disease activity/presence of malignancy within 5 years, except for adequately treated basal cell carcinoma of the skin, cervical dysplasia, or carcinoma in situ of the skin or the cervix
* Known human immunodeficiency virus (HIV) or Hepatitis B/C (HBV/HCV) infection
* Has a history of hospitalization for any psychiatric disorder, or any suicide attempt in the 2 years prior to Screening
* Is actively abusing alcohol or drugs or has a history of alcohol or drug abuse during the 6 months prior to Screening
* Is being treated for hypothyroidism, but the dose of medication has not been stable for at least 3 months at the time of Screening
* Is a pregnant, breast-feeding, or lactating woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Actual)
Dates: Start 2013-04; Primary Completion 2014-03 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (94):
- United States (46):
  - Alabama Clinical Therapeutics, Birmingham, Alabama
  - G and L Research, LLC, Foley, Alabama
  - Adobe Gastroenterology Research, LLC, Tucson, Arizona
  - Skyline Research LLC, Cerritos, California
  - GW Research, Inc., Chula Vista, California
  - Paradigm Clinical, Inc., Garden Grove, California
  - Providence Clinical Research, North Hollywood, California
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - Pulmonary Associates of Brandon, Brandon, Florida
  - In Vivo Clinical Research, Inc., Hialeah, Florida
  - Medsearch Professional Group, Inc., Hialeah, Florida
  - The Community Research of South Florida, Hialeah, Florida
  - Center for Gastrointestinal Disorders, Hollywood, Florida
  - Nature Coast Clinical Research, LLC, Inverness, Florida
  - Gastroenterology and Hepatology Associates, Jacksonville, Florida
  - Jupiter Research Inc., Jupiter, Florida
  - Center for Advanced Gastroenterology, Maitland, Florida
  - Advanced Pharma CR, LLC, Miami, Florida
  - Research Institute of South Florida, Miami, Florida
  - Gastroenterology Group of Naples, Naples, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Georgia Clinical Research, Snellville, Georgia
  - Elite Clinical Trials, Inc., Blackfoot, Idaho
  - MediSphere Medical Research Center, LLC, Evansville, Indiana
  - MidAtlantic Medical Research Centers, Philip J. Bean Medical Center, Hollywood, Maryland
  - Boston Clinical Trials, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Midwest Gastroenterology Partners, Lee's Summit, Missouri
  - Advanced Biomedical Research of America, Las Vegas, Nevada
  - ActivMed Practices and Research, Inc., Newington, New Hampshire
  - HOSC, Inc., Brooklyn, New York
  - North American Partners in Pain Management, Valley Stream, New York
  - Carolina Digestive Health Associates, PA, Davidson, North Carolina
  - Cumberland Research Associates, LLC, Fayetteville, North Carolina
  - Gastroenterology Research Consultants of Greater Cincinnati, Cincinnati, Ohio
  - Hometown Urgent Care and Occupational Health, Groveport, Ohio
  - Oklahoma Foundation for Digestive Research, Oklahoma City, Oklahoma
  - Clinical Trials Research Services, LLC, Pittsburgh, Pennsylvania
  - Mainline Gastroenterology Associates, Souderton, Pennsylvania
  - ClinSearch, Chattanooga, Tennessee
  - Memphis Gastroenterology Group, PC, Germantown, Tennessee
  - KRK Medical Research, Dallas, Texas
  - Research Across America, Dallas, Texas
  - Pioneer Research Solutions, Inc., Houston, Texas
  - Pioneer Research Solutions, Inc., Sugar Land, Texas
  - Northwest Gastroenterology Associates, Bellevue, Washington
- Belgium (3):
  - Cliniques Universitaires Saint Luc, Brussels, Brussels Capital
  - Huisartspraktijk Jaak Mortelmans, Ham
  - Universitair Ziekenhuis Leuven, Leuven
- Brazil (3):
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Faculdade de Medicina do ABC, Sant André, São Paulo
  - Escola Paulista de Medicina, Universidade Federal de São Paulo, São Paulo, São Paulo
- Canada (5):
  - John Buhler Research Center, Winnipeg, Manitoba
  - Maritime Medical Research Center, Bathurst, New Brunswick
  - Prime Health Clinical Research Organization, Toronto, Ontario
  - Alpha Clinical Research LLC, Québec, Quebec
  - Rhodin Recherche Clinique, DrummondvilleQC
- Czechia (3):
  - Derma Plus s.r.o., České Budějovice
  - Gastroenterologie, s. r. o., Hradec Králové
  - Nemocnice Valasske Mezirici a.s., Gastroenterologicka ambulance, Valašské Meziříčí
- Germany (9):
  - Klinikum der Universität München-Großhadern, München, Bavaria
  - Israelitisches Krankenhaus Hamburg, Hamburg, Hamburg
  - Synexus Clinical Research GmbH, Frankfurt am Main, Hesse
  - Elbe Klinikum Stade - Buxtehude GmbH, Stade, Lower Saxony
  - Synexus Clinical Research GmbH, Bochum, North Rhine-Westphalia
  - Synexus Clinical Research GmbH, Leipzig, Saxony
  - Emovis GmbH, Berlin, State of Berlin
  - Synexus Clinical Research GmbH, Berlin, State of Berlin
  - Universitätsklinik Charité, Campus Mitte, Berlin, State of Berlin
- Israel (6):
  - Soroka University Medical Center, Beersheba
  - Bnai Zion Medical Center, Haifa
  - Hadassah Medical Organization, Ein Kerem, Jerusalem
  - Kaplan Medical Center, Rehovot
  - Sheba Medical Center, Tel Litwinsky
  - Assaf Harofeh Medical Centre, Ẕerifin
- Poland (5):
  - Szpital Wojewódzki w Opolu, Opole, Opole Voivodeship
  - Centrum Medyczne sw. Lukasza Sp. z o.o., Częstochowa, Silesian Voivodeship
  - Neuro-Care NZOZ, Katowice, Silesian Voivodeship
  - Pomorski Uniwersytet Medyczny, Szczecin, West Pomeranian Voivodeship
  - SPZOZ Uniwersytecki Szpital Kliniczny nr 5 im. Gen. Dyw. B. Szareckiego, Uniwersytetu Medycznego, Lódz, Łódź Voivodeship
- South Africa (8):
  - Global Clinical Trials, Port Elizabeth, Eastern Cape
  - Boanerges Clinical Research, Bloemfontein, Free State
  - Synexus Clinical Research SA, Pretoria, Gauteng
  - Parklands Medical Centre, Durban, KwaZulu-Natal
  - Boland Ethical Research Group, Worcester, Western Cape
  - The Memory Centre, Johannesburg
  - Langeberg Clinical Trials, Kraaifontein
  - Newtown Clinical Research Centre, Newtown
- United Kingdom (6):
  - Synexus Midlands Clinical Research Centre, Birmingham, England
  - County Durham and Darlington NHS Foundation Trust, Durham, England
  - Synexus Manchester Clinical Research Centre, Manchester, England
  - Tayside University Hospitals NHS Trust, Ninewells Hospital and Medical School, Dundee, Scotland
  - Synexus Wales Clinical Research Centre, Cardiff, Wales
  - Nottingham University Hospitals NHS Trust, Nottingham

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The trial included a 4-week Screening Period and a 2-week Pretreatment Period prior to patient randomization to a 26-week Treatment Period. A total of 909 patients were screened in the trial and of these 533 patients were excluded due to screening failure.
Groups:
- EBX 10: Elobixibat 10 mg/day was administered orally in a tablet form starting from Baseline visit till End of the Treatment (EoT) visit.
- EBX 5: Elobixibat 5 mg/day as administered orally in a tablet form starting from Baseline visit till EoT visit.
- PLCBO: Placebo was administered orally in a tablet form starting from Baseline visit till EoT visit.
Period: Overall Study
Arm/Group | EBX 10 | EBX 5 | PLCBO
Started | 126 (Randomized patients.) | 126 (Randomized patients.) | 124 (Randomized patients.)
Safety Analysis Set | 125 (1 patient withdrew consent before getting the treatment.) | 126 | 124
Completed | 52 | 46 | 48
Not Completed | 74 | 80 | 76
Not completed — Adverse Event | 11 | 9 | 2
Not completed — Physician Decision | 0 | 2 | 1
Not completed — Protocol Violation | 2 | 1 | 0
Not completed — Lost to Follow-up | 1 | 2 | 2
Not completed — Withdrawal by Subject | 12 | 11 | 11
Not completed — Patient's substantial non-compliance | 1 | 1 | 6
Not completed — Trial terminated by Sponsor | 47 | 53 | 51
Not completed — Others | 0 | 1 | 3

BASELINE CHARACTERISTICS:
Population: Intention-to-treat population
Groups:
- EBX 10: Elobixibat 10 mg/day was administered orally in a tablet form starting from Baseline visit till EoT visit.
- EBX 5: Elobixibat 5 mg/day was administered orally in a tablet form starting from Baseline visit till EoT visit.
- Total: Total of all reporting groups
Arm/Group | EBX 10 | EBX 5 | PLCBO | Total
Number analyzed (Participants) | 126 | 126 | 124 | 376
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 110 | 113 | 112 | 335
  >=65 years | 16 | 13 | 12 | 41
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.0 (14.3) | 45.8 (14.1) | 46.1 (14.4) | 46.6 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 107 | 103 | 314
  Male | 22 | 19 | 21 | 62
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 32 | 28 | 86
  Not Hispanic or Latino | 100 | 94 | 96 | 290
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 2
  Asian | 2 | 4 | 7 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 28 | 23 | 29 | 80
  White | 95 | 97 | 87 | 279
  More than one race | 0 | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 6 | 6 | 5 | 17
  Czech Republic | 2 | 2 | 2 | 6
  Belgium | 2 | 2 | 2 | 6
  United States | 73 | 78 | 77 | 228
  Poland | 2 | 1 | 0 | 3
  United Kingdom | 12 | 10 | 9 | 31
  South Africa | 14 | 11 | 14 | 39
  Germany | 15 | 16 | 15 | 46
Weekly number of CSBM [Mean (Standard Deviation); unit: CSBM per week] — CSBM was defined as a spontaneous (occurring without laxative within the preceding 24 hours, including no rescue medication within the preceding 24 hours) bowel movement (as interpreted by the patient, with a beginning and an end, including single or multiple stools), accompanied by a patient reported sense of complete evacuation ('complete').
  Baseline value for the number of CSBM per week was defined as the average of the numbers of CSBM per week for over the 2-week Pretreatment Period.
  CSBM per week | 0.36 (0.66) | 0.44 (0.75) | 0.54 (0.82) | 0.45 (0.75)
Weekly number of SBM [Mean (Standard Deviation); unit: SBM per week] — SBM was defined as a bowel movement that occurs in the absence of a laxative use or manual disimpaction.
  Baseline value for the number of SBM was defined as the average of the numbers of SBM per week for over the 2-week Pretreatment Period.
  SBM per week | 2.20 (1.34) | 2.13 (1.27) | 2.31 (1.43) | 2.21 (1.35)

OUTCOME MEASURES:

1. Primary Outcome: Overall Complete Spontaneous Bowel Movement (CSBM) Response
Description: This outcome measured the percentage of patients who were CSBM responders. A CSBM responder was defined as a patient with ≥3 CSBMs per week and an increase of ≥1 CSBM per week from Baseline, for at least 9 of the 12 weeks in the 12-week Treatment Period, including at least 3 weeks during Weeks 9-12.
Time Frame: During the first 12 weeks
Population: Intention-to-treat (ITT) analysis set consisted of all randomized (as planned) patients.
Measure: Number; unit: Percentage of patients
Arm/Group | EBX 10 | EBX 5 | PLCBO
Number analyzed (Participants) | 126 | 126 | 124
Percentage of patients | 15.9 | 23.0 | 12.1

2. Secondary Outcome: Occurrence of CSBM Response
Description: This outcome measured the percentage of patients who had a CSBM within 24 hours after the first dose of treatment. A CSBM was defined as a spontaneous (occurring without laxative within the preceding 24 hours, including no rescue medication within the preceding 24 hours) bowel movement (as interpreted by the patient, with a beginning and an end, including single or multiple stools), accompanied by a patient reported sense of complete evacuation ('complete').
Time Frame: Within the first 24 hours of treatment initiation
Population: The ITT analysis set consisted of all randomized (as planned) patients was used for assessment.
Measure: Number; unit: Percentage of patients
Arm/Group | EBX 10 | EBX 5 | PLCBO
Number analyzed (Participants) | 126 | 126 | 124
Percentage of patients | 20.6 | 24.6 | 12.1

3. Secondary Outcome: Change From Baseline in Weekly Frequency of Spontaneous Bowel Movements (SBMs)
Description: The change from Baseline for the continuous variable was estimated using a repeated measures analysis of covariance (ANCOVA) model.
Time Frame: From Baseline (2-week Pretreatment Period) to overall first 12-weeks of Treatment Period
Population: The ITT analysis set consisted of all randomized (as planned) patients.
Measure: Least Squares Mean (95% Confidence Interval); unit: SBM per week
Arm/Group | EBX 10 | EBX 5 | PLCBO
Number analyzed (Participants) | 126 | 126 | 124
SBM per week | 2.04 [1.64 to 2.44] | 2.44 [2.04 to 2.84] | 1.55 [1.15 to 1.95]

4. Secondary Outcome: Change From Baseline in Weekly Stool Consistency of SBMs
Description: The stool consistency is measured using the seven-point ordinal Bristol Stool Form Scale (BSFS) score. The BSFS classifies human stool into seven types and points them accordingly.
  Type 1: Separate hard lumps, like nuts (hard to pass) Type 2: Sausage-shaped, but lumpy Type 3: Like a sausage but with cracks on its surface Type 4: Like a sausage or snake, smooth and soft Type 5: Soft blobs with clear cut edges (passed easily) Type 6: Fluffy pieces with ragged edges, a mushy stool Type 7: Watery, no solid pieces, entirely liquid Types 1 and 2 indicate constipation, with 3 and 4 represents the ideal stool form (especially the latter), and 5, 6 and 7 tends towards diarrhoea .
  For a given assessment week, the weekly stool consistency was defined as the sum of non-missing stool consistency score for SBMs during that week divided by the number of non-missing stool consistency score for SBMs during that week. The parameter was analysed using repeated measures ANCOVA model.
Time Frame: From Baseline (2-week Pretreatment Period) to overall first 12-weeks of Treatment Period
Population: The ITT analysis set consisted of all randomized (as planned) patients.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on BSFS
Arm/Group | EBX 10 | EBX 5 | PLCBO
Number analyzed (Participants) | 126 | 126 | 124
Units on BSFS | 1.41 [1.24 to 1.58] | 1.35 [1.18 to 1.52] | 0.83 [0.66 to 1.00]

5. Secondary Outcome: Total Patient Assessment of Constipation - Quality of Life (PAC-QOL) Score Responder
Description: This outcome measured the percentage of patients who were PAC-QOL score responder at 12-week of Treatment Period. A PAC-QOL score responder was defined as a patient with ≥50% reduction in total PAC-QOL score from Baseline at Week 12.
  PAC-QOL is a 28-item questionnaire for psychometric assessment of disease-specific quality of life. The questionnaire is based on 5-point Likert scale; ranging from 0 [none of the time or not at all] to 4 [all of the time or extremely]). A lower score indicates a better Quality of Life. The PAC-QOL questionnaire is developed specifically for patients with constipation.
  Total PAC-QOL score was averaged from the individual item score.
Time Frame: At 12 weeks
Population: The ITT analysis set consisted of all randomized (as planned) patients.
Measure: Number; unit: Percentage of patients
Arm/Group | EBX 10 | EBX 5 | PLCBO
Number analyzed (Participants) | 126 | 126 | 124
Percentage of patients | 34.1 | 33.3 | 25.8

6. Secondary Outcome: Change From Baseline in Weekly Degree of Straining of SBMs
Description: The degree of straining was measured using the five-point ordinal scale (1=Not at all, 2=A little bit, 3=A moderate amount, 4=A great deal, and 5=An extreme amount).
  For a given assessment week, the weekly degree of straining was defined as the sum of non-missing straining score for SBMs during that week divided by the number of non-missing straining score for SBMs during that week. The parameter was analysed using repeated measures ANCOVA model.
Time Frame: From Baseline (2-week Pretreatment Period) to overall first 12-weeks of Treatment Period
Population: The ITT analysis set consisted of all randomized (as planned) patients.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | EBX 10 | EBX 5 | PLCBO
Number analyzed (Participants) | 126 | 126 | 124
Units on a scale | -1.01 [-1.15 to -0.88] | -1.04 [-1.17 to -0.91] | -0.91 [-1.05 to -0.78]

7. Secondary Outcome: Change From Baseline in Weekly Abdominal Bloating Score
Description: The abdominal bloating score was measured using the five-point ordinal scale (1=None, 2=Mild, 3=Moderate, 4=Severe, and 5=Very severe).
  For a given assessment week, the weekly abdominal bloating score was defined as the sum of non-missing abdominal bloating score for SBMs during that week divided by the number of non-missing abdominal bloating score for SBMs during that week. The parameter was analysed using repeated measures ANCOVA model.
Time Frame: From Baseline (2-week Pretreatment Period) to overall first 12-weeks of Treatment Period
Population: The ITT analysis set consisted of all randomized (as planned) patients.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | EBX 10 | EBX 5 | PLCBO
Number analyzed (Participants) | 126 | 126 | 124
Units on a scale | -0.49 [-0.61 to -0.38] | -0.52 [-0.63 to -0.40] | -0.35 [-0.47 to -0.24]

8. Secondary Outcome: Change From Baseline in Weekly Abdominal Discomfort Score
Description: The abdominal discomfort score was measured using the five-point ordinal scale (1=None, 2=Mild, 3=Moderate, 4=Severe, and 5=Very severe).
  For a given assessment week, the weekly abdominal discomfort score was defined as the sum of non-missing abdominal discomfort score for SBMs during that week divided by the number of non-missing abdominal discomfort score for SBMs during that week. The parameter was analysed using repeated measures ANCOVA model.
Time Frame: From Baseline (2-week Pretreatment Period) to overall first 12-weeks of Treatment Period
Population: The ITT analysis set consisted of all randomized (as planned) patients.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | EBX 10 | EBX 5 | PLCBO
Number analyzed (Participants) | 126 | 126 | 124
Units on a scale | -0.43 [-0.54 to -0.32] | -0.46 [-0.57 to -0.35] | -0.38 [-0.49 to -0.27]

ADVERSE EVENTS:
Time Frame: 34 weeks
Description: The Investigator monitored the condition of the patient and recorded all AEs throughout the trial from the time of obtaining informed consent until the last visit (i.e. the end of the follow-up period, as applicable) in the AEs Log . Information on AEs was collected at each trial visit.
Arm/Group | EBX 10 | EBX 5 | PLCBO
Serious Adverse Events (participants affected / at risk) | 3/125 | 3/126 | 1/124
Other Adverse Events (participants affected / at risk) | 42/125 | 28/126 | 23/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EBX 10 (N=125) | EBX 5 (N=126) | PLCBO (N=124)
Glaucoma (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EBX 10 (N=125) | EBX 5 (N=126) | PLCBO (N=124)
Abdominal pain (Gastrointestinal disorders) | 18 (22) | 6 (6) | 7 (11)
Diarrhoea (Gastrointestinal disorders) | 11 (21) | 9 (14) | 3 (4)
Nasopharyngitis (Infections and infestations) | 10 (10) | 7 (7) | 11 (12)
Urinary tract infection (Infections and infestations) | 7 (8) | 5 (6) | 3 (3)
Headache (Nervous system disorders) | 6 (7) | 7 (7) | 5 (5)

LIMITATIONS AND CAVEATS:
Due to the early termination of the study, outcomes were presented only for descriptive purposes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.